CLINICAL TRIAL: NCT00632541
Title: A Phase II Study of Combined VEGF Inhibitor (Bevacizumab + Sorafenib) in Patients With Metastatic Breast Cancer: Hoosier Oncology Group BRE06-109
Brief Title: A Phase II Study of Bevacizumab + Sorafenib in Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Significant Toxicities Experienced
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Genentech, Inc. (Industry); Bayer (Industry); Amgen (Industry)
Responsible Party: Principal Investigator, Robin Zon, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRE06-109
Record Dates: First submitted 2008-02-28; First posted 2008-03-10 (Estimated); Results first posted 2016-01-07 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Sorafenib; Bevacizumab; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm A (Experimental): Sorafenib 200mg po daily, Bevacizumab 5mg/kg every other week, 1 Cycle = 4 weeks. Imaging every third cycle
  Interventions: Drug: Sorafenib; Drug: Bevacizumab; Other: Imaging

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 200mg po daily
Drug: Bevacizumab — Bevacizumab 5mg/kg every other week
  1 Cycle = 4 weeks
Other: Imaging — Imaging every third cycle

SUMMARY:
Prior clinical trials involving bevacizumab and sorafenib have demonstrated single agent activity in previously treated advanced breast cancer. This trial will test combined VEGF inhibition with sorafenib and bevacizumab in less heavily pre-treated patients with advanced breast cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Sorafenib 200mg po daily Bevacizumab 5mg/kg every other week

1 Cycle = 4 weeks Imaging every third cycle

Acceptable toxicity and non-PD = Protocol therapy will continue Un-acceptable toxicity or PD = Protocol therapy will be discontinued

ECOG Performance Status 0-1

Life Expectancy: at least 12 weeks

Hematopoietic:

* Platelets > 100 K/mm3
* Absolute neutrophil count (ANC) > 1.5 K/mm3
* Hemoglobin > 10 g/dL

Hepatic:

* Total Bilirubin < 1.5 x ULN
* Aspartate aminotransferase (AST, SGOT) < 2 x ULN (up to 5 x ULN in patients with known liver involvement)

Renal:

* Creatinine < 1.5 x ULN
* No proteinuria as demonstrated by either Urine protein:creatinine (UPC) ratio < 1.0 or Urine dipstick for proteinuria < 2+

Cardiovascular:

* No known myocardial infarction, unstable angina, > grade II New York Heart Association (NYHA) classification, congestive heart failure, uncontrolled hypertension defined as SBP >150 or DBP >100, > grade II peripheral vascular disease or significant vascular disease (e.g. aortic aneurysm, aortic dissection) within 12 months prior to being registered for protocol therapy.
* No uncontrolled or clinically significant arrhythmia. NOTE: Controlled atrial fibrillation is allowed.
* LVEF ≥ LLN by MUGA or ECHO as obtained within 28 days prior to being registered for protocol therapy.

Pulmonary:

* No pulmonary hemorrhage/bleeding event ≥ CTCAE grade 2 within 28 days prior to being registered for protocol therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of breast cancer with evidence of metastatic disease. NOTE: Patients with Her-2 positive (3+ by IHC or gene amplification by FISH) are eligible only if they have had prior trastuzumab therapy.
* Must have measurable or non-measurable lesions as defined by the Response Evaluation Criteria in Solid Tumors (RECIST).
* Two or fewer prior chemotherapy regimens in any disease setting. NOTE: All adjuvant and neoadjuvant chemotherapy will be considered one regimen. NOTE: Prior hormonal therapy for metastatic disease is allowed. NOTE: Prior radiation therapy is allowed as long as the irradiated area is not the only source of evaluable disease.
* Age > 18 years at the time of consent.
* Written informed consent and HIPAA authorization for release of personal health information.
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 8 weeks after treatment discontinuation.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy.
* Ability to comply with study and/or follow-up procedures.

Exclusion Criteria:

* No prior therapy with bevacizumab, sorafenib or any other known VEGF inhibitors.
* No known hypersensitivity to any component of the study drugs.
* No other forms of cancer therapy including radiation, chemotherapy and hormonal therapy within 21 days prior to being registered for protocol therapy.
* No history or radiologic evidence of CNS metastases including previously treated, resected, or asymptomatic brain lesions or leptominigeal involvement. A head CT or MRI must be obtained within 28 days prior to being registered for protocol therapy.
* No other participation in another clinical drug study within 28 days prior to being registered for protocol therapy.
* No known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C
* No major surgical procedure within 28 days prior to being registered for protocol therapy or anticipation of need for major surgical procedure during the course of the study. Placement of a vascular access device and breast biopsy will not be considered major surgery.
* No minor surgical procedure within 7 days prior to being registered for protocol therapy.
* No known history of cerebrovascular disease including TIA, stroke or subarachnoid hemorrhage.
* No known history of ischemic bowel.
* No known history of deep venous thrombosis or pulmonary embolism.
* No history of hypertensive crisis or hypertensive encephalopathy.
* No non-healing wound or fracture.
* No active infection requiring parenteral antibiotics.
* No other hemorrhage/bleeding event ≥ CTCAE grade 3 within 28 days prior to being registered for protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin T Zon, M.D., Principal Investigator — Hoosier Oncology Group, Inc.; Kathy Miller, M.D., Principal Investigator — Hoosier Oncology Group, Inc.
Locations (10):
- United States (10):
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Ireland Cancer Center - University Hospitals of Cleveland, Cleveland, Ohio

REFERENCES:
- [Result] Mina LA, Yu M, Johnson C, Burkhardt C, Miller KD, Zon R. A phase II study of combined VEGF inhibitor (bevacizumab+sorafenib) in patients with metastatic breast cancer: Hoosier Oncology Group Study BRE06-109. Invest New Drugs. 2013 Oct;31(5):1307-10. doi: 10.1007/s10637-013-9976-1. Epub 2013 Jun 28. PMID 23812905
- See also: Hoosier Cancer Research Network Homepage — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm A: Sorafenib 200mg po daily, Bevacizumab 5mg/kg every other week. 1 Cycle = 4 weeks. Imaging every third cycle.
Period: Overall Study
Arm/Group | Single Arm A
Started | 18 (18 subjects were accrued to the study)
Completed | 11
Not Completed | 7
Not completed — Adverse Event | 7

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm A
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 56 [33 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
ECOG Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group performance status - scale from zero to five, 0 - fully functional, 5 - dead.
  participants
    ECOG = 0 | 13
    ECOG = 1 | 5
Breast Cancer Subtype [Number; unit: participants] — Estrogen receptor (ER), progesterone receptor (PR), human epidermal receptor 2 (HER2) status - positive (+), negative (-).
  participants
    ER-/PR-/HER2- | 8
    ER-/PR-/HER2+ | 1
    ER+/PR-/HER2- | 4
    ER+/PR+/HER2- | 3
    ER+/PR+/HER2 unknown | 2
Prior Chemotherapy Regimens [Number; unit: participants] — Prior chemotherapy regimens - 0 - regimens, 1-2 regimens
  participants
    Prior Chemotherapy Regimens - 0 | 1
    Prior Chemotherapy Regimens 1-2 | 17
Prior Hormone Therapy [Number; unit: participants] — Prior hormone therapy; none or any.
  participants
    No Prior Hormone Therapy | 9
    Prior Hormone Therapy | 9
Prior Radiation Therapy [Number; unit: participants] — Prior Radiation Therapy; none, any
  participants
    No Prior Radiation Therapy | 7
    Prior Radiation Therapy | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: The primary objective was to assess the Progression-Free Survival of sorafenib combined with bevacizumab in patients with metastatic breast cancer. Progression is defined by RECIST as a 20% increase in the sum of the longest diameters of target measurable lesions over the smallest sum observed (over baseline if no decrease during therapy) or by the appearance of a new lesion.
Time Frame: From the start of the treatment until the criteria for disease progression is met (or death occurs) maximum of 24 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Single Arm A: Sorafenib 200mg po daily, Bevacizumab 5mg/kg every other week, 1 Cycle = 4 weeks. Imaging every third cycle
  Sorafenib: Sorafenib 200mg po daily
  Bevacizumab: Bevacizumab 5mg/kg every other week
  1 Cycle = 4 weeks
  Imaging: Imaging every third cycle
Arm/Group | Single Arm A
Number analyzed (Participants) | 18
months | 2.8 [1.8 to 6.1]

2. Secondary Outcome: Assess the Clinical Benefit Response: the Proportion of Patients With Clinical Benefit (CR+PR+SD > 6 Months Duration) Will be Assessed at the Completion of the Study.
Time Frame: 6 months
Population: Data for this secondary objective was not collected or analyzed
Arm/Group | Single Arm A
Number analyzed (Participants) | 0

3. Secondary Outcome: Assess the Overall Response Rate.
Time Frame: 24 months
Population: Data for this secondary objective was not collected or analyzed.
Arm/Group | Single Arm A
Number analyzed (Participants) | 0

4. Secondary Outcome: Determine the Adverse Event Profile of Sorafenib Combined With Bevacizumab in This Patient Population.
Time Frame: 24 months
Population: Data for this secondary objective was not collected or analyzed.
Arm/Group | Single Arm A
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Single Arm A
Serious Adverse Events (participants affected / at risk) | 4/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm A (N=18)
ASCITES (NON-MALIGNANT) (Gastrointestinal disorders) | 1 (1)
DEATH NOT ASSOCIATED WITH CTCAE TERM / DISEASE PROGRESSION NOS (General disorders) | 1 (1)
NEUROPATHY: SENSORY (Nervous system disorders) | 1 (1)
PAIN / CHEST WALL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm A (N=18)
ALKALINE PHOSPHATASE (Investigations) | 1 (1)
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 1 (1)
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Immune system disorders) | 1 (1)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 1 (1)
ANOREXIA (Gastrointestinal disorders) | 5 (6)
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 1 (1)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 3 (4)
AUDITORY/EAR - OTHER (SPECIFY, __) (Ear and labyrinth disorders) | 1 (1)
CARDIAC ARRHYTHMIA - OTHER (SPECIFY, __) (Cardiac disorders) | 1 (1)
CARDIAC GENERAL - OTHER (SPECIFY, __) (Cardiac disorders) | 1 (1)
CONFUSION (Nervous system disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 8 (9)
COUGH (Respiratory, thoracic and mediastinal disorders) | 9 (10)
DEHYDRATION (Gastrointestinal disorders) | 1 (1)
DERMATOLOGY/SKIN - OTHER (SPECIFY, __) (Skin and subcutaneous tissue disorders) | 5 (7)
DIARRHEA (Gastrointestinal disorders) | 6 (9)
DIZZINESS (Nervous system disorders) | 2 (2)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 6 (7)
EDEMA: LIMB (Blood and lymphatic system disorders) | 2 (2)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 15 (21)
FLU-LIKE SYNDROME (General disorders) | 1 (1)
GASTROINTESTINAL - OTHER (SPECIFY, __) (Gastrointestinal disorders) | 1 (1)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 1 (2)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 1 (1)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 4 (5)
HEMORRHAGE, GI / RECTUM (Gastrointestinal disorders) | 2 (2)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / NOSE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HOT FLASHES/FLUSHES (Endocrine disorders) | 5 (5)
HYPERTENSION (Cardiac disorders) | 15 (18)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / ABDOMEN NOS (Infections and infestations) | 1 (1)
INSOMNIA (General disorders) | 4 (4)
LYMPHATICS - OTHER (SPECIFY, __) (Blood and lymphatic system disorders) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 1 (1)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 4 (4)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Surgical and medical procedures) | 4 (4)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ORAL CAVITY (Gastrointestinal disorders) | 3 (4)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-UPPER (Musculoskeletal and connective tissue disorders) | 1 (4)
NAUSEA (Gastrointestinal disorders) | 8 (13)
NEUROPATHY: SENSORY (Nervous system disorders) | 5 (7)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 2 (5)
PAIN / BACK (General disorders) | 4 (5)
PAIN / CARDIAC/HEART (Cardiac disorders) | 1 (2)
PAIN / CHEST WALL (Respiratory, thoracic and mediastinal disorders) | 2 (3)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 1 (3)
PAIN / DENTAL/TEETH/PERIDONTAL (Gastrointestinal disorders) | 1 (1)
PAIN / EXTERNAL EAR (Ear and labyrinth disorders) | 1 (1)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 7 (8)
PAIN / HEAD/HEADACHE (General disorders) | 6 (6)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 4 (6)
PAIN / MUSCLE (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN / NECK (General disorders) | 2 (3)
PAIN / ORAL CAVITY (Gastrointestinal disorders) | 1 (1)
PAIN / PAIN NOS (General disorders) | 1 (2)
PAIN / PELVIS (General disorders) | 1 (1)
PAIN / RECTUM (Gastrointestinal disorders) | 2 (2)
PAIN / TUMOR PAIN (General disorders) | 1 (1)
PAIN - OTHER (SPECIFY, __) (General disorders) | 5 (7)
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PROTEINURIA (Investigations) | 2 (3)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 2 (2)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1)
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 4 (6)
RENAL/GENITOURINARY - OTHER (SPECIFY, __) (Renal and urinary disorders) | 1 (1)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 2 (2)
TINNITUS (Ear and labyrinth disorders) | 2 (2)
URINARY RETENTION (INCLUDING NEUROGENIC BLADDER) (Renal and urinary disorders) | 1 (1)
VOICE CHANGES/DYSARTHRIA (E.G., HOARSENESS, LOSS OR ALTERATION IN VOICE, LARYNGITIS) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
VOMITING (Gastrointestinal disorders) | 4 (4)
WEIGHT LOSS (General disorders) | 3 (5)
WOUND COMPLICATION, NON-INFECTIOUS (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to a poor safety profile as well as the lack of significant efficacy of this combination over bevacizumab alone in the short followup period where it was evaluated. Therefore, secondary objectives were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No